CLINICAL TRIAL: NCT02571777
Title: A Multicenter, Randomized, 52-week, Double-blind, Parallelgroup, Active Controlled Study to Compare the Efficacy and Safety of QVM149 With QMF149 in Patients With Asthma
Brief Title: Study to Compare the Efficacy and Safety of QVM149 With QMF149 in Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVM149B2302; 2015-002899-25 (EudraCT Number)
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Asthma; QVM149; QMF149
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- QVM149 150/50/160 µg o.d. (Experimental): QVM149 150/50/160 μg (indacaterol acetate/glycopyrronium/mometasone furoate) once daily (o.d.) delivered via Concept1 device
  Interventions: Drug: QVM149 150/50/160
- QVM149 150/50/80 µg o.d. (Experimental): QVM149 150/50/80 μg (indacaterol acetate/glycopyrronium/mometasone furoate) once daily (o.d.) delivered via Concept1 device
  Interventions: Drug: QVM149 150/50/80
- QMF149 150/320 µg o.d. (Active Comparator): QMF149 150/320 μg (indacaterol acetate/mometasone furoate) once daily (o.d.) delivered via Concept1 device
  Interventions: Drug: QMF149 150/320
- QMF149 150/160 µg o.d. (Active Comparator): QMF149 150/160 μg (indacaterol acetate/mometasone furoate) once daily (o.d.) delivered via Concept1 device
  Interventions: Drug: QMF149 150/160
- Salmeterol/fluticasone 50/500 μg b.i.d. (Active Comparator): Salmeterol xinafoate /fluticasone propionate 50/500 μg twice daily (b.i.d.) delivered via Accuhaler®
  Interventions: Drug: salmeterol/fluticasone

INTERVENTIONS:
Drug: QVM149 150/50/160
  Arms: QVM149 150/50/160 µg o.d.
Drug: QVM149 150/50/80
  Arms: QVM149 150/50/80 µg o.d.
Drug: QMF149 150/320
  Arms: QMF149 150/320 µg o.d.
Drug: QMF149 150/160
  Arms: QMF149 150/160 µg o.d.
Drug: salmeterol/fluticasone
  Arms: Salmeterol/fluticasone 50/500 μg b.i.d.

SUMMARY:
The purpose of the trial was to evaluate the efficacy and safety of two different doses of QVM149 (QVM149 150/50/80 μg and QVM149 150/50/160 μg via Concept1) over two respective QMF149 doses (QMF149 150/160 μg and QMF149 150/320) μg via Concept1 in poorly controlled asthmatics as determined by pulmonary function testing and effects on asthma control.

DETAILED DESCRIPTION:
This study used a 52-week treatment, randomized, double-blind, double-dummy, parallel-group design. A total of 3092 asthma patients were randomized into the 5 treatment groups with a randomization ratio of 1:1:1:1:1 (approximately 617 patients per treatment group): QVM149 150/50/80 μg once daily (o.d.), QVM149 150/50/160 μg o.d., QMF149 150/160 μg o.d. and QMF149 150/320 μg o.d., all delivered via the Concept1 device, and salmeterol/fluticasone 50/500 μg twice daily (b.i.d.) delivered via Accuhaler. The 52 week treatment period was followed by a 30-day Follow-up.

The primary objective of this study was to demonstrate superiority of either QVM149 150/50/80 μg o.d. to QMF149 150/160 μg o.d. or QVM149 150/50/160 μg o.d. to QMF149 150/320 μg o.d in terms of trough Forced Expiratory Volume in One Second (Trough FEV1) (FEV1) at Week 26, all delivered via Concept1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of asthma, (GINA 2015) for a period of at least 1 year prior to Visit 1 (Screening).
* Patients who have used medium or high dose of ICS/LABA combinations for asthma for at least 3 months and at stable medium or high doses of ICS/LABA for at least 1 month prior to Visit 1.
* Patients must be symptomatic at screening despite treatment with mid or high stable doses of ICS/LABA. Patients with ACQ-7 score ≥ 1.5 at Visit 101 and at Visit 102 (before randomization).
* Patients with documented history of at least one asthma exacerbation which required medical care from a physician, ER visit (or local equivalent structure) or hospitalization in the 12 months prior to Visit 1, and required systemic corticosteroid treatment.
* Pre-bronchodilator FEV1 of < 80 % of the predicted normal value for the patient according to ATS/ERS guidelines after withholding bronchodilators at both visits 101 and 102.
* Withholding period of bronchodilators prior to spirometry: SABA for ≥ 6 hrs, Twice daily LABA (or FDC of ICS/LABA) for ≥ 12 hrs, Once daily LABA (or FDC of ICS/LABA) for ≥ 24 hrs, SAMA for ≥ 8 hrs, Short acting xanthines for 12 hrs, Long acting xanthines for 24 hrs, .
* Washout period of each drug should be kept as close as possible as above and should not be longer. If longer washout period is needed due to scheduling issues, please contact Novartis Medical monitor.
* A one-time repeat of percentage predicated FEV1 (Pre-bronchodilator) at Visit 101 and/or Visit 102 is allowed in an ad-hoc visit. Repeat of Visit 101 spirometry should be done in an ad-hoc visit to be scheduled on a date that would provide sufficient time to receive confirmation from the spirometry data central reviewer of the validity of the assessment before randomization. Run-in medication should be dispensed once spirometry assessment met inclusion criteria (ATS/ERS quality criteria, FEV1 % predicted normal value, and reversibility) as per equipment
* A one-time rescreen is allowed in case the patient fails to meet the criteria at the repeat, provided the patient returned to the required treatment as per inclusion criteria 4
* Patients who demonstrate an increase in FEV1 of 12% and 200 mL within 30 minutes after administration of 400 µg salbutamol/360 µg albuterol (or equivalent dose) at Visit 101.All patients must perform a reversibility test at Visit 101. If reversibility is not demonstrated at Visit 101 then one of the following criteria need to be met.
* Reversibility should be repeated once.
* Patients may be permitted to enter the study with historical evidence of reversibility that was performed according to ATS/ERS guidelines within 2 years prior to Visit 1.
* Alternatively, patients may be permitted to enter the study with a historical positive bronchoprovocation test that was performed within 2 years prior to Visit 1. If reversibility is not demonstrated at Visit 101 (or after repeated assessment in an ad-hoc visit) and historical evidence of reversibility/bronchoprovocation is not available (or was not performed according to the ATS/ERS guidelines patients must be screen failed
* Spacer devices are permitted during reversibility testing only. The Investigator or delegate may decide whether or not to use a spacer for the reversibility testing

Exclusion Criteria:

* Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of Visit 1 (Screening). If patients experience an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit between Visit 1 and Visit 102 they may be re-screened 6 weeks after recovery from the exacerbation.
* Patients who have ever required intubation for a severe asthma attack/exacerbation.
* Patients who have a clinical condition which is likely to be worsened by ICS administration (e.g. glaucoma, cataract and fragility fractures) who are according to investigator's medical judgment at risk participating in the study.
* Patients treated with a LAMA for asthma within 3 months prior Visit 1 (Screening).
* Patients with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia (BPH) or bladder-neck obstruction or severe renal impairment or urinary retention. BPH patients who are stable on treatment can be considered).
* Patients who have had a respiratory tract infection or asthma worsening as determined by investigator within 4 weeks prior to Visit 1 (Screening) or between Visit 1 and Visit 102. Patients may be re-screened 4 weeks after recovery from their respiratory tract infection or asthma worsening.
* Patients with evidence upon visual inspection (laboratory culture is not required) of clinically significant (in the opinion of investigator) oropharyngeal candidiasis at Visit 102 or earlier, with or without treatment. Patients may be re-screened once their candidiasis has been treated and has resolved.
* Patients with any chronic conditions affecting the upper respiratory tract (e.g. chronic sinusitis) which in the opinion of the investigator may interfere with the study evaluation or optimal participation in the study.
* Patients with a history of chronic lung diseases other than asthma, including (but not limited to) chronic obstructive pulmonary disease, sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Patients with Type I diabetes or uncontrolled Type II diabetes.
* Patients who, either in the judgment of the investigator or the responsible Novartis personnel, have a clinically significant condition such as (but not limited to) unstable ischemic heart disease, New York Heart Association (NYHA) Class III/IV left ventricular failure arrhythmia, uncontrolled hypertension, cerebrovascular disease, psychiatric disease, neurodegenerative diseases, or other neurological disease, uncontrolled hypo- and hyperthyroidism and other autoimmune diseases, hypokalemia, hyperadrenergic state, or ophthalmologic disorder or patients with a medical condition that might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study.
* Patients with paroxysmal (e.g., intermittent) atrial fibrillation are excluded. Patients with persistent atrial fibrillation as defined by continuous atrial fibrillation for at least 6 months and controlled with a rate control strategy (i.e., selective beta blockers, calcium channel blocker, pacemaker placement, digoxin or ablation therapy) for at least 6 months may be considered for inclusion. In such patients, atrial fibrillation must be present at the run-in visit (Visit 101) with a resting ventricular rate < 100/min. At Visit 101 the atrial fibrillation must be confirmed by central reading.
* Patients with a history of myocardial infarction (this should be confirmed clinically by the investigator) within the previous 12 months.
* Concomitant use of agents known to prolong the QT interval unless it can be permanently discontinued for the duration of study
* Patients with a history of long QT syndrome or whose QTc measured at Visit 101 (Fridericia method) is prolonged (> 450 msec for males and > 460 msec for females) and confirmed by a central assessor (these patients should not be rescreened).
* Patients with a history of hypersensitivity to lactose, any of the study drugs or to similar drugs within the class including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof.
* Patients who have not achieved an acceptable spirometry result at Visit 101 in accordance with ATS/ERS criteria for acceptability and repeatability. A one-time repeat spirometry is allowed in an ad-hoc visit scheduled as close as possible from the first attempt (but not on the same day) if the spirometry did not qualify due to ATS/ERS criteria at Visit 101 and/or Visit 102. If the patient fails the repeat assessment, the patient may be rescreened once, provided the patient returns to the required treatment as per inclusion criteria 4.
* Patients unable to use the Concept1 dry powder inhaler, Accuhaler or a metered dose inhaler. Spacer devices are not permitted.
* History of alcohol or other substance abuse.
* Patients with a known history of non-compliance to medication or who were unable or unwilling to complete a patient diary or who are unable or unwilling to use Electronic Peak Flow with e-diary device.
* Patients who do not maintain regular day/night, waking/sleeping cycles (e.g., night shift workers).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3092 (Actual)
Dates: Start 2015-12-08 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (320):
- Argentina (19):
  - Novartis Investigative Site, Bahía Blanca, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Nueve de Julio, Buenos Aires
  - Novartis Investigative Site, San Nicolás de los Arroyos, Buenos Aires
  - Novartis Investigative Site, Vicente López, Buenos Aires
  - Novartis Investigative Site, Villa María, Córdoba Province
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, Godoy Cruz, Mendoza Province
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Paraná
  - Novartis Investigative Site, Santa Fe
- Austria (4):
  - Novartis Investigative Site, Bludenz
  - Novartis Investigative Site, Feldbach
  - Novartis Investigative Site, Feldkirch
  - Novartis Investigative Site, Grieskirchen
- Belgium (10):
  - Novartis Investigative Site, Gosselies, BEL
  - Novartis Investigative Site, Hasselt, BEL
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Braine L Alleud Waterloo
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Éghezée
  - Novartis Investigative Site, Lebbeke
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Malmedy
- Bulgaria (4):
  - Novartis Investigative Site, Plovdiv, BGR
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
- Canada (9):
  - Novartis Investigative Site, Sherwood Park, Alberta
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
  - Novartis Investigative Site, Victoriaville, Quebec
  - Novartis Investigative Site, Québec
- Chile (4):
  - Novartis Investigative Site, Curicó, Maule Region
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
  - Novartis Investigative Site, Valparaíso, TX
  - Novartis Investigative Site, Santiago
- China (11):
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (4):
  - Novartis Investigative Site, Bogota DC
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Floridablanca
  - Novartis Investigative Site, Medellín
- Croatia (4):
  - Novartis Investigative Site, Zagreb, HRV
  - Novartis Investigative Site, Petrinja
  - Novartis Investigative Site, Zadar
  - Novartis Investigative Site, Zagreb
- Denmark (2):
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Hvidovre
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Jyväskylä, Finland
- Novartis Investigative Site, Montpellier, Herault, France
- Germany (23):
  - Novartis Investigative Site, Bochum, North Rhine-Westphalia
  - Novartis Investigative Site, Koblenz, North Rhine-Westphalia
  - Novartis Investigative Site, Cottbus, Saxony
  - Novartis Investigative Site, Geesthacht, Schleswig-Holstein
  - Novartis Investigative Site, Annaberg-Buchholz
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mittweida
  - Novartis Investigative Site, Neu-Isenburg
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Witten
- Greece (4):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Hungary (16):
  - Novartis Investigative Site, Budaörs, HUN
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Eger, HUN
  - Novartis Investigative Site, Kapuvár, HUN
  - Novartis Investigative Site, Püspökladány, HUN
  - Novartis Investigative Site, Tata, HUN
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Mátészalka
  - Novartis Investigative Site, Nyíregyháza
  - Novartis Investigative Site, Szarvas
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szigetszentmiklós
  - Novartis Investigative Site, Szigetvár
- India (29):
  - Novartis Investigative Site, Guntur, Andhra Pradesh
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Vijayawada, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Patna, Bihar
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Hubli, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Cherthala, Kerala
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Mohali, Punjab
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Kanpur, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, Kolkata, West Bengal
- Ireland (2):
  - Novartis Investigative Site, Wilton, Cork
  - Novartis Investigative Site, Dublin
- Israel (7):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Giborim, Holon
- Italy (10):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Ancona
  - Novartis Investigative Site, Messina
  - Novartis Investigative Site, Pordenone
  - Novartis Investigative Site, Roma
- Japan (20):
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Tomakomai, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Naka-gun, Ibaraki
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokkaichi, Mie-ken
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Tokyo, Shibuya Ku
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Kokubunji, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo
- Novartis Investigative Site, Amman, JOR, Jordan
- Latvia (9):
  - Novartis Investigative Site, Balvi, LVA
  - Novartis Investigative Site, Bauska, LVA
  - Novartis Investigative Site, Daugavpils, LVA
  - Novartis Investigative Site, Jūrmala, LVA
  - Novartis Investigative Site, Rēzekne, LVA
  - Novartis Investigative Site, Riga, LVA
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Lebanon (3):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Lithuania (7):
  - Novartis Investigative Site, Vilnius, LTU
  - Novartis Investigative Site, Kaunas, LT
  - Novartis Investigative Site, Vilnius, LT
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Vilnius
- Mexico (6):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Culiacan, State of Mexico
  - Novartis Investigative Site, Oaxaca City
  - Novartis Investigative Site, Veracruz
- Netherlands (9):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Harderwijk
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Helmond
  - Novartis Investigative Site, Hengelo
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Zutphen
- Peru (5):
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
  - Novartis Investigative Site, Lima
- Philippines (5):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Bulacan
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (12):
  - Novartis Investigative Site, Aleksandrow Odzki, Poland
  - Novartis Investigative Site, Ksawerów, POL
  - Novartis Investigative Site, Wejherowo, POL
  - Novartis Investigative Site, Bielsko-Biala
  - Novartis Investigative Site, Elblag
  - Novartis Investigative Site, Inowrocław
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zawadzkie
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Romania (11):
  - Novartis Investigative Site, Craiova, ROM
  - Novartis Investigative Site, Deva, ROM
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Arad
  - Novartis Investigative Site, Bacau
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Constanța
  - Novartis Investigative Site, Deva
  - Novartis Investigative Site, Piteşti
- Russia (24):
  - Novartis Investigative Site, Ulyanovsk, Russian Federation
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Pskov
  - Novartis Investigative Site, Pyatigorsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Vladikavkaz
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Vsevolozhsk
  - Novartis Investigative Site, Yaroslavl
- Slovakia (10):
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Liptovský Mikuláš
  - Novartis Investigative Site, Poprad
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Spišská Nová Ves
  - Novartis Investigative Site, Trenčín
  - Novartis Investigative Site, Zvolen
  - Novartis Investigative Site, Žilina
- South Africa (4):
  - Novartis Investigative Site, Berea, Durban
  - Novartis Investigative Site, Durban, KwaZulu-Natal
  - Novartis Investigative Site, Kempton Park, ZAF
  - Novartis Investigative Site, Cape Town
- Spain (12):
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Esparraguera, Barcelona
  - Novartis Investigative Site, Laredo, Cantabria
  - Novartis Investigative Site, Vila-real, Castellon
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, León
  - Novartis Investigative Site, Zaragoza
- Sweden (2):
  - Novartis Investigative Site, Lidingö
  - Novartis Investigative Site, Stockholm
- Novartis Investigative Site, Gossau, Switzerland
- Thailand (4):
  - Novartis Investigative Site, Muang, Changwat Nonthaburi
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (3):
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Wiltshire
- Vietnam (3):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] van Zyl-Smit RN, Kerstjens HAM, Maspero J, Tanase AM, Lawrence D, Mezzi K, D'Andrea P, Chapman KR. Triple Therapy with Mometasone/Indacaterol/Glycopyrronium or Doubling the ICS/LABA Dose in GINA Step 4: IRIDIUM Analyses. Pulm Ther. 2023 Sep;9(3):395-409. doi: 10.1007/s41030-023-00234-y. Epub 2023 Aug 1. PMID 37526856
- [Derived] Kostikas K, Maspero JF, Chapman KR, Mezzi K, Jaumont X, Lawrence D, van Zyl-Smit R. Efficacy of mometasone/indacaterol/glycopyrronium in patients with inadequately controlled asthma with respect to baseline eosinophil count: Post hoc analysis of IRIDIUM study. Respir Med. 2023 Oct;217:107334. doi: 10.1016/j.rmed.2023.107334. Epub 2023 Jun 29. PMID 37392789
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Chapman K, van Zyl-Smit R, Maspero J, Kerstjens HAM, Gon Y, Hosoe M, Tanase AM, Pethe A, Shu X, D'Andrea P. One time a day mometasone/indacaterol fixed-dose combination versus two times a day fluticasone/salmeterol in patients with inadequately controlled asthma: pooled analysis from PALLADIUM and IRIDIUM studies. BMJ Open Respir Res. 2021 Aug;8(1):e000819. doi: 10.1136/bmjresp-2020-000819. PMID 34452934
- [Derived] Kerstjens HAM, Maspero J, Chapman KR, van Zyl-Smit RN, Hosoe M, Tanase AM, Lavecchia C, Pethe A, Shu X, D'Andrea P; IRIDIUM trial investigators. Once-daily, single-inhaler mometasone-indacaterol-glycopyrronium versus mometasone-indacaterol or twice-daily fluticasone-salmeterol in patients with inadequately controlled asthma (IRIDIUM): a randomised, double-blind, controlled phase 3 study. Lancet Respir Med. 2020 Oct;8(10):1000-1012. doi: 10.1016/S2213-2600(20)30190-9. Epub 2020 Jul 9. PMID 32653074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 415 investigative sites in 41 countries
Pre-assignment Details: 4851 participants were screened of which 3092 participants were randomized to 1 of the 5 treatment groups with a randomization ratio of 1:1:1:1:1.
Period: Overall Study
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Started (All patients who were assigned a randomization number) | 619 | 620 | 618 | 617 | 618
Full Analysis Set (FAS) (All patients in the randomization set who received at least one dose of study medication) | 615 | 616 | 611 | 607 | 612
Safety Set (SAF) (All patients who received at least one dose of study medication whether or not being randomized) | 616 | 617 | 613 | 608 | 618
Completed | 580 | 582 | 577 | 580 | 582
Not Completed | 39 | 38 | 41 | 37 | 36
Not completed — Subject/guardian decision | 34 | 26 | 26 | 25 | 27
Not completed — Protocol Deviation | 2 | 3 | 4 | 8 | 4
Not completed — Death | 1 | 1 | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0 | 1
Not completed — Physician Decision | 1 | 7 | 5 | 2 | 4
Not completed — Pregnancy | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set (RAN) consisted of all participants who were assigned a randomization number, regardless of whether or not they actually received study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d. | Total
Number analyzed (Participants) | 619 | 620 | 618 | 617 | 618 | 3092
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (12.91) | 52.4 (12.71) | 52.0 (12.81) | 51.8 (12.86) | 52.9 (12.23) | 52.2 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 381 | 362 | 380 | 378 | 417 | 1918
  Male | 238 | 258 | 238 | 239 | 201 | 1174
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 456 | 458 | 453 | 452 | 468 | 2287
  Black | 4 | 5 | 3 | 4 | 1 | 17
  Asian | 139 | 133 | 133 | 135 | 131 | 671
  Native American | 7 | 8 | 8 | 4 | 5 | 32
  Unknown | 0 | 0 | 0 | 1 | 0 | 1
  Other | 13 | 16 | 21 | 21 | 13 | 84

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in 1 Second (Trough FEV1) of QVM149 Versus QMF149 at Week 26
Description: Trough FEV1 was assessed by performing spirometric assessment. It is defined as average of the two FEV1 measurements taken 23 hr 15 min and 23 hr 45 min post-evening dose. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
  The primary endpoint considered the following 2 comparison groups:
  * QVM149 150/50/80 μg o.d. compared with QMF149 150/160 μg o.d. both delivered via Concept1
  * QVM149 150/50/160 μg o.d. compared with QMF149 150/320 μg o.d. both delivered via Concept1.
Time Frame: 26 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: litre (L)
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 614 | 614 | 606 | 602 | 607
litre (L) | 2.050 (0.0128) | 2.029 (0.0129) | 1.984 (0.0129) | 1.953 (0.0130) | 1.930 (0.0131)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p < 0.001, Mixed Model for Repeated Measures (MMRM); LS Mean = 0.065, 95% CI 2-sided [0.031 to 0.099], Standard Error of Mean 0.0176
Statistical Analysis 2: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.076, 95% CI 2-sided [0.041 to 0.111], Standard Error of Mean 0.0176

2. Secondary Outcome: Asthma Control Questionnaire (ACQ-7) at Week 26 and Week 52
Description: The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 on airway calibre (FEV1 % predicted). All 7 questions of the ACQ-7 were equally weighted. Items 1-5 were scored along a 7-point response scale, where 0 = totally controlled and 6 = severely uncontrolled. Item 6 is scored between 0 = no rescue medication and 6 = More than 16 puffs/inhalations most days. The 7th item was scored by the investigator based on the FEV1 % predicted from the masterscope at the site (i.e., Score = 0 means > 95% of predicted FEV1, 1 = 90 - 95%, 2 = 80 - 89%, 3 = 70 - 79%, 4 = 60 - 69%, 5 = 50 - 59%, and Score = 6 means < 50% of predicted FEV1). The ACQ-7 total score reported below was calculated as the mean of scores of all 7 items and ranged between 0 and 6, with higher scores indicating worse asthma symptom control.
Time Frame: 26 weeks, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 607 | 595 | 596 | 598 | 599
Score on a scale
  Week 26: number analyzed (Participants) | 566 | 559 | 562 | 559 | 562
  Week 26 | 1.542 (0.0329) | 1.543 (0.0330) | 1.528 (0.0329) | 1.614 (0.0331) | 1.628 (0.0329)
  Week 52: number analyzed (Participants) | 552 | 537 | 547 | 536 | 547
  Week 52 | 1.406 (0.0334) | 1.535 (0.0337) | 1.465 (0.0335) | 1.545 (0.0338) | 1.527 (0.0335)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 26; Test type: Superiority; p = 0.729, MMRM; LS Mean = 0.014, 95% CI 2-sided [-0.066 to 0.094], Standard Error of Mean 0.0406
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.034, MMRM; LS Mean = -0.086, 95% CI 2-sided [-0.165 to -0.006], Standard Error of Mean 0.0404
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 26; Test type: Superiority; p = 0.085, MMRM; LS Mean = -0.071, 95% CI 2-sided [-0.151 to 0.010], Standard Error of Mean 0.0409
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.038, MMRM; LS Mean = -0.084, 95% CI 2-sided [-0.164 to -0.005], Standard Error of Mean 0.0406
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 52; Test type: Superiority; p = 0.157, MMRM; LS Mean = -0.059, 95% CI 2-sided [-0.140 to 0.023], Standard Error of Mean 0.0415
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.003, MMRM; LS Mean = -0.121, 95% CI 2-sided [-0.202 to -0.040], Standard Error of Mean 0.0414
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 52; Test type: Superiority; p = 0.814, MMRM; LS Mean = -0.010, 95% CI 2-sided [-0.092 to 0.072], Standard Error of Mean 0.0420
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.845, MMRM; LS Mean = 0.008, 95% CI 2-sided [-0.073 to 0.090], Standard Error of Mean 0.0416

3. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (Trough FEV1) of QVM149 Versus Salmeterol/Fluticasone at Week 26
Description: Trough FEV1 was assessed by performing spirometric assessment. It is defined as average of the two FEV1 measurements taken 23 hr 15 min and 23 hr 45 min post-evening dose. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
  This secondary endpoint considered the following 2 comparison groups:
  * QVM149 150/50/80 μg o.d. via Concept1 compared with salmeterol/fluticasone 50/500 μg b.i.d. via Accuhaler®
  * QVM149 150/50/160 μg o.d. via Concept 1 compared with salmeterol/fluticasone 50/500 μg b.i.d. via Accuhaler®
Time Frame: 26 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: litre (L)
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 614 | 614 | 606 | 602 | 607
litre (L) | 2.050 (0.0128) | 2.029 (0.0129) | 1.984 (0.0129) | 1.953 (0.0130) | 1.930 (0.0131)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.119, 95% CI 2-sided [0.085 to 0.154], Standard Error of Mean 0.0177
Statistical Analysis 2: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.099, 95% CI 2-sided [0.064 to 0.133], Standard Error of Mean 0.0177

4. Secondary Outcome: Trough FEV1 at Week 52
Description: Trough FEV1 was assessed by performing spirometric assessment. It is defined as average of the two FEV1 measurements taken 23 hr 15 min and 23 hr 45 min post-evening dose. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Time Frame: 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: litre (L)
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 614 | 614 | 606 | 602 | 607
litre (L) | 2.050 (0.0129) | 1.992 (0.0130) | 1.965 (0.0130) | 1.930 (0.0130) | 1.905 (0.0132)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.086, 95% CI 2-sided [0.051 to 0.120], Standard Error of Mean 0.0176
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.145, 95% CI 2-sided [0.111 to 0.180], Standard Error of Mean 0.0178
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.062, 95% CI 2-sided [0.027 to 0.096], Standard Error of Mean 0.0178
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.087, 95% CI 2-sided [0.052 to 0.122], Standard Error of Mean 0.0179

5. Secondary Outcome: Pre-dose Forced Vital Capacity (FVC) at Week 4 and Week 12
Description: Pre-dose FVC is defined as average of the two FVC measurements taken 45 min and 15 min pre evening dose. It was assessed by performing spirometric assessment. FVC is the total amount of air exhaled during the FEV test.
Time Frame: 4 weeks, 12 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: litre (L)
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 606 | 594 | 592 | 596 | 598
litre (L)
  Week 4: number analyzed (Participants) | 598 | 573 | 573 | 579 | 577
  Week 4 | 3.091 (0.0161) | 3.059 (0.0163) | 3.018 (0.0163) | 3.020 (0.0163) | 2.952 (0.0163)
  Week 12: number analyzed (Participants) | 580 | 569 | 573 | 562 | 568
  Week 12 | 3.067 (0.0162) | 3.065 (0.0164) | 3.011 (0.0163) | 3.014 (0.0164) | 2.965 (0.0163)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.073, 95% CI 2-sided [0.030 to 0.116], Standard Error of Mean 0.0218
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.139, 95% CI 2-sided [0.096 to 0.181], Standard Error of Mean 0.0217
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 4; Test type: Superiority; p = 0.074, MMRM; LS Mean = 0.039, 95% CI 2-sided [-0.004 to 0.082], Standard Error of Mean 0.0220
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.108, 95% CI 2-sided [0.065 to 0.150], Standard Error of Mean 0.0219
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 12; Test type: Superiority; p = 0.010, MMRM; LS Mean = 0.056, 95% CI 2-sided [0.014 to 0.099], Standard Error of Mean 0.0219
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 12; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.102, 95% CI 2-sided [0.059 to 0.145], Standard Error of Mean 0.0218
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 12; Test type: Superiority; p = 0.022, MMRM; LS Mean = 0.050, 95% CI 2-sided [0.007 to 0.094], Standard Error of Mean 0.0221
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 12; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.099, 95% CI 2-sided [0.056 to 0.142], Standard Error of Mean 0.0220

6. Secondary Outcome: Trough Forced Expiratory Flow (FEF) Between 25% and 75% of FVC (FEF25-75) at 52 Weeks
Description: FEF is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration. Trough FEF25-75% is defined as average of the two FEF25-75% measurements taken 23 hr 15 min and 23 hr 45 min post-evening dose. It was assessed by performing spirometric assessment.
Time Frame: Up to Week 52
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: L/s
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 614 | 614 | 606 | 602 | 607
L/s | 1.354 (0.0190) | 1.263 (0.0192) | 1.260 (0.0191) | 1.214 (0.0192) | 1.207 (0.0194)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.095, 95% CI 2-sided [0.045 to 0.145], Standard Error of Mean 0.0254
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.147, 95% CI 2-sided [0.097 to 0.198], Standard Error of Mean 0.0256
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.057, MMRM; LS Mean = 0.049, 95% CI 2-sided [-0.001 to 0.099], Standard Error of Mean 0.0256
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.029, MMRM; LS Mean = 0.056, 95% CI 2-sided [0.006 to 0.107], Standard Error of Mean 0.0258

7. Secondary Outcome: Change From Baseline in Morning and Evening Peak Expiratory Flow Rate (PEF) Over 26 and 52 Weeks of Treatment
Description: PEF is a person's maximum speed of expiration. All the participants were instructed to record PEF twice daily using a mini Peak Flow Meter device, once in the morning (before taking the morning dose) and once approximately 12 h later in the evening (before taking the evening dose) at home. At each timepoint, the participant was instructed to perform 3 consecutive manoeuvres within 10 minutes. These PEF values were captured in the e-PEF/diary. The best of 3 values were used.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 596 | 584 | 581 | 584 | 586
L/min
  Week 26 - Mean morning PEF: number analyzed (Participants) | 596 | 583 | 581 | 584 | 584
  Week 26 - Mean morning PEF | 47.7 (1.93) | 40.5 (1.95) | 29.5 (1.95) | 25.6 (1.95) | 12.5 (1.95)
  Week 26 - Mean evening PEF: number analyzed (Participants) | 594 | 584 | 580 | 578 | 577
  Week 26 - Mean evening PEF | 39.6 (1.87) | 34.7 (1.88) | 22.8 (1.88) | 20.6 (1.89) | 10.4 (1.89)
  Week 52 - Mean morning PEF: number analyzed (Participants) | 596 | 584 | 581 | 583 | 586
  Week 52 - Mean morning PEF | 47.5 (2.03) | 41.2 (2.05) | 28.8 (2.05) | 25.6 (2.06) | 12.7 (2.05)
  Week 52 - Mean evening PEF: number analyzed (Participants) | 593 | 577 | 578 | 576 | 578
  Week 52 - Mean evening PEF | 38.7 (1.97) | 35.0 (1.99) | 21.2 (1.99) | 20.1 (2.00) | 9.2 (1.99)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 26 - Mean morning PEF; Test type: Superiority; p < 0.001, Linear Mixed Model (LMM); LS Mean = 18.2, 95% CI 2-sided [13.2 to 23.3], Standard Error of Mean 2.59
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26 - Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 35.3, 95% CI 2-sided [30.2 to 40.3], Standard Error of Mean 2.58
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 26 - Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 14.9, 95% CI 2-sided [9.8 to 20.0], Standard Error of Mean 2.61
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26 - Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 28.0, 95% CI 2-sided [22.9 to 33.1], Standard Error of Mean 2.60
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 26 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 16.8, 95% CI 2-sided [11.8 to 21.7], Standard Error of Mean 2.53
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 29.1, 95% CI 2-sided [24.2 to 34.1], Standard Error of Mean 2.53
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 26 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 14.1, 95% CI 2-sided [9.1 to 19.1], Standard Error of Mean 2.55
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 24.3, 95% CI 2-sided [19.3 to 29.3], Standard Error of Mean 2.54
Statistical Analysis 9: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 52 - Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 18.7, 95% CI 2-sided [13.4 to 24.1], Standard Error of Mean 2.72
Statistical Analysis 10: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52 - Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 34.8, 95% CI 2-sided [29.5 to 40.1], Standard Error of Mean 2.70
Statistical Analysis 11: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 52 - Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 15.6, 95% CI 2-sided [10.2 to 20.9], Standard Error of Mean 2.74
Statistical Analysis 12: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52 - Mean morning PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 28.5, 95% CI 2-sided [23.2 to 33.8], Standard Error of Mean 2.72
Statistical Analysis 13: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 52 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 17.5, 95% CI 2-sided [12.3 to 22.8], Standard Error of Mean 2.66
Statistical Analysis 14: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 29.5, 95% CI 2-sided [24.2 to 34.7], Standard Error of Mean 2.66
Statistical Analysis 15: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 52 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 15.0, 95% CI 2-sided [9.7 to 20.2], Standard Error of Mean 2.69
Statistical Analysis 16: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52 - Mean evening PEF; Test type: Superiority; p < 0.001, LMM; LS Mean = 25.8, 95% CI 2-sided [20.5 to 31.0], Standard Error of Mean 2.68

8. Secondary Outcome: Change From Baseline in Percentage of Asthma Symptom-free Days Over 52 Weeks
Description: All participants were provided with an electronic diary (e-Diary) to record clinical symptoms. They were instructed to routinely complete the e-Diary twice daily at the same time each morning and again approximately 12 hours later in the evening. The e-Diary was reviewed at each visit until study completion. Asthma symptoms free days are days with no daytime symptoms, no night-time awakenings and no symptoms on awakening. The daytime asthma symptom score was based on the daily e-diary recordings by participants with respect to shortness of breath, wheeze, cough, chest tightness, and impact on usual daily activities due to symptoms.
Time Frame: Baseline, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 566 | 552 | 559 | 554 | 558
Percentage of days | 22.4 (1.35) | 18.0 (1.36) | 22.2 (1.36) | 18.0 (1.37) | 18.9 (1.36)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p = 0.907, LMM; LS Mean = 0.2, 95% CI 2-sided [-3.3 to 3.8], Standard Error of Mean 1.81
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.055, LMM; LS Mean = 3.5, 95% CI 2-sided [-0.1 to 7.0], Standard Error of Mean 1.81
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.997, LMM; LS Mean = 0.0, 95% CI 2-sided [-3.6 to 3.6], Standard Error of Mean 1.83
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.606, LMM; LS Mean = -0.9, 95% CI 2-sided [-4.5 to 2.6], Standard Error of Mean 1.82

9. Secondary Outcome: Change From Baseline in Percentage of Days With no Daytime Symptoms Over 52 Weeks
Description: All participants were provided with an electronic diary (e-Diary) to record clinical symptoms. They were instructed to routinely complete the e-Diary twice daily at the same time each morning and again approximately 12 hours later in the evening. The e-Diary was reviewed at each visit until study completion. For days with no daytime symptoms, all 5 evening questions must have a score = 0 with respect to shortness of breath, wheeze, cough, chest tightness and impact on usual daily activities due to symptoms, each with scores from 0 (no problems) to 4 (very severe problems).
Time Frame: Baseline, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 594 | 577 | 579 | 579 | 578
Percentage of days | 22.5 (1.32) | 17.9 (1.34) | 21.8 (1.33) | 18.0 (1.34) | 18.8 (1.34)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p = 0.712, LMM; LS Mean = 0.7, 95% CI 2-sided [-2.8 to 4.2], Standard Error of Mean 1.78
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.038, LMM; LS Mean = 3.7, 95% CI 2-sided [0.2 to 7.2], Standard Error of Mean 1.78
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.943, LMM; LS Mean = -0.1, 95% CI 2-sided [-3.7 to 3.4], Standard Error of Mean 1.80
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.612, LMM; LS Mean = -0.9, 95% CI 2-sided [-4.4 to 2.6], Standard Error of Mean 1.79

10. Secondary Outcome: Change From Baseline in Percentage of Nights With no Night-time Awakenings Over 52 Weeks
Description: All participants were provided with an electronic diary (e-Diary) to record clinical symptoms. They were instructed to routinely complete the e-Diary twice daily at the same time each morning and again approximately 12 hours later in the evening. The e-Diary was reviewed at each visit until study completion. The question asked for nights with no night-time awakenings was "How did you sleep last night?" had to be answered with "I did not wake up because of any breathing problems" with scores from 0 (no problem)-4 (very severe problems).
Time Frame: Baseline, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 599 | 584 | 582 | 584 | 586
Percentage of days | 18.0 (1.11) | 17.6 (1.12) | 18.4 (1.13) | 16.1 (1.13) | 16.9 (1.12)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p = 0.809, LMM; LS Mean = -0.4, 95% CI 2-sided [-3.3 to 2.6], Standard Error of Mean 1.51
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.467, LMM; LS Mean = 1.1, 95% CI 2-sided [-1.9 to 4.0], Standard Error of Mean 1.50
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.318, LMM; LS Mean = 1.5, 95% CI 2-sided [-1.5 to 4.5], Standard Error of Mean 1.52
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.640, LMM; LS Mean = 0.7, 95% CI 2-sided [-2.3 to 3.7], Standard Error of Mean 1.51

11. Secondary Outcome: Change From Baseline in Percentage of Mornings With no Symptoms on Rising Over 52 Weeks
Description: as for outcome 10
Time Frame: Baseline, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 599 | 584 | 582 | 584 | 586
Percentage of days | 19.5 (1.33) | 18.5 (1.35) | 19.9 (1.35) | 15.5 (1.35) | 15.6 (1.34)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p = 0.814, LMM; LS Mean = -0.4, 95% CI 2-sided [-4.0 to 3.2], Standard Error of Mean 1.83
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.036, LMM; LS Mean = 3.8, 95% CI 2-sided [0.2 to 7.4], Standard Error of Mean 1.83
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.098, LMM; LS Mean = 3.1, 95% CI 2-sided [-0.6 to 6.7], Standard Error of Mean 1.84
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.118, LMM; LS Mean = 2.9, 95% CI 2-sided [-0.7 to 6.5], Standard Error of Mean 1.84

12. Secondary Outcome: Change From Baseline in Percentage of Days Without Rescue Medication Use Over 26 and 52 Weeks
Description: Percentage of days without rescue medication usage (100 μg salbutamol/90 μg albuterol via metered-dose inhaler) as recorded by e-diary over 26 and 52 weeks of treatment.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 590 | 577 | 578 | 580 | 579
Percentage of days
  Week 26 | 22.5 (1.32) | 19.5 (1.33) | 23.3 (1.33) | 18.2 (1.33) | 19.6 (1.33)
  Week 52: number analyzed (Participants) | 583 | 574 | 576 | 576 | 578
  Week 52 | 25.0 (1.36) | 21.9 (1.36) | 24.9 (1.36) | 20.8 (1.37) | 21.8 (1.36)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 26; Test type: Superiority; p = 0.645, LMM; LS Mean = -0.8, 95% CI 2-sided [-4.2 to 2.6], Standard Error of Mean 1.74
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.095, LMM; LS Mean = 2.9, 95% CI 2-sided [-0.5 to 6.3], Standard Error of Mean 1.73
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 26; Test type: Superiority; p = 0.460, LMM; LS Mean = 1.3, 95% CI 2-sided [-2.1 to 4.7], Standard Error of Mean 1.75
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.971, LMM; LS Mean = -0.1, 95% CI 2-sided [-3.5 to 3.4], Standard Error of Mean 1.75
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 52; Test type: Superiority; p = 0.963, LMM; LS Mean = 0.1, 95% CI 2-sided [-3.4 to 3.6], Standard Error of Mean 1.78
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.075, LMM; LS Mean = 3.2, 95% CI 2-sided [-0.3 to 6.6], Standard Error of Mean 1.77
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 52; Test type: Superiority; p = 0.517, LMM; LS Mean = 1.2, 95% CI 2-sided [-2.3 to 4.7], Standard Error of Mean 1.79
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.956, LMM; LS Mean = 0.1, 95% CI 2-sided [-3.4 to 3.6], Standard Error of Mean 1.78

13. Secondary Outcome: Percentage of Patients Achieving the Minimal Clinically Important Difference (MCID) ACQ ≥ 0.5 at Week 26 and Week 52
Description: Change from baseline in ACQ-7 scores of ≤ 0.5 was defined as minimal clinically important difference and were considered clinically meaningful. The ACQ-7 measured asthma symptom control and consists of 7 items: 5 on symptom assessment, 1 on rescue bronchodilator use and 1 on airway calibre (FEV1 % predicted). All 7 questions of the ACQ-7 were equally weighted. Items 1-5 were scored along a 7-point response scale, where 0 = totally controlled and 6 = severely uncontrolled. Item 6 is scored between 0 = no rescue medication and 6 = More than 16 puffs/inhalations most days. The 7th item was scored by the investigator based on the FEV1 % predicted from the masterscope at the site (i.e., Score = 0 means > 95% of predicted FEV1, 1 = 90 - 95%, 2 = 80 - 89%, 3 = 70 - 79%, 4 = 60 - 69%, 5 = 50 - 59%, and Score = 6 means < 50% of predicted FEV1). The total score was calculated as the mean of all questions.
Time Frame: 26 weeks, 52 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
Percentage of participants
  Week 26: number analyzed (Participants) | 566 | 559 | 562 | 559 | 562
  Week 26 | 71.2 | 71.7 | 74.2 | 70.7 | 67.4
  Week 52: number analyzed (Participants) | 552 | 537 | 547 | 536 | 547
  Week 52 | 78.8 | 72.8 | 77.9 | 73.1 | 72.8
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 26; Test type: Superiority; p = 0.535, Logistic regression model; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.70 to 1.20]
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.151, Logistic regression model; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.93 to 1.57]
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 26; Test type: Superiority; p = 0.380, Logistic regression model; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.86 to 1.48]
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.172, Logistic regression model; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.92 to 1.57]
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 52; Test type: Superiority; p = 0.510, Logistic regression model; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.83 to 1.47]
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.017, Logistic regression model; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.06 to 1.86]
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 52; Test type: Superiority; p = 0.744, Logistic regression model; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.79 to 1.38]
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.922, Logistic regression model; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.75 to 1.29]

14. Secondary Outcome: Time to First Hospitalization for Asthma Exacerbation
Description: Time from start of treatment until the first event (hospitalization for asthma exacerbation) or censoring. Patients without the event were considered as censored at the date of last treatment + 1 day. For patients having the event, the start date of the hospitalization was considered to calculate the time to event (i.e., the number of days from start of treatment up to the event start date).
Time Frame: 52 weeks on average, up to 416 days
Population: FAS
Measure: Median (Full Range); unit: days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
days | 367.0 [2 to 416] | 367.0 [2 to 396] | 367.0 [1 to 411] | 367.0 [1 to 408] | 367.0 [1 to 416]
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p = 0.371, Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.27 to 1.63]
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.996, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.37 to 2.66]
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.145, Regression, Cox; Hazard Ratio (HR) = 1.89, 95% CI 2-sided [0.80 to 4.47]
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.150, Regression, Cox; Hazard Ratio (HR) = 1.88, 95% CI 2-sided [0.80 to 4.43]

15. Secondary Outcome: Time to First Asthma Exacerbation by Exacerbation Category
Description: Time from start of treatment until the first event (asthma exacerbation) or censoring. Patients without the event were considered as censored at the date of last treatment + 1 day. For patients having the event, the start date of the exacerbation was considered to calculate the time to event (i.e., the number of days from start of treatment up to the event start date).
  The exacerbation categories were: All (mild, moderate and severe), combination of moderate or severe and severe.
Time Frame: 52 weeks on average, up to 416 days
Population: FAS
Measure: Median (Full Range); unit: days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
days
  Moderate or severe asthma exacerbation | 366.0 [2 to 416] | 366.0 [2 to 396] | 366.0 [1 to 411] | 365.0 [1 to 387] | 365.0 [1 to 416]
  Severe asthma exacerbation | 366.0 [2 to 416] | 366.0 [2 to 396] | 366.0 [1 to 411] | 366.0 [1 to 389] | 366.0 [1 to 416]
  All (mild, moderate or severe) asthma exacerbation | 363.0 [2 to 416] | 364.0 [2 to 396] | 361.0 [1 to 411] | 360.0 [1 to 384] | 278.0 [1 to 416]
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.523, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.77 to 1.15]
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.58 to 0.84]
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.164, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.06]
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.005, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.63 to 0.92]
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Severe asthma exacerbation; Test type: Superiority; p = 0.476, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.72 to 1.16]
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Severe asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.54 to 0.85]
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Severe asthma exacerbation; Test type: Superiority; p = 0.243, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.70 to 1.09]
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Severe asthma exacerbation; Test type: Superiority; p = 0.027, Regression, Cox; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.63 to 0.97]
Statistical Analysis 9: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.497, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.79 to 1.12]
Statistical Analysis 10: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.60 to 0.84]
Statistical Analysis 11: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.126, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.73 to 1.04]
Statistical Analysis 12: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.61 to 0.85]

16. Secondary Outcome: Annual Rate of Asthma Exacerbations by Exacerbation Category
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: 52 weeks
Population: FAS
Measure: Mean (95% Confidence Interval); unit: Exacerbations per year
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
Exacerbations per year
  Moderate or severe asthma exacerbation: number analyzed (Participants) | 615 | 615 | 611 | 607 | 612
  Moderate or severe asthma exacerbation | 0.46 [0.39 to 0.54] | 0.58 [0.50 to 0.67] | 0.54 [0.47 to 0.63] | 0.67 [0.58 to 0.77] | 0.72 [0.63 to 0.82]
  Severe asthma exacerbation: number analyzed (Participants) | 615 | 615 | 611 | 607 | 612
  Severe asthma exacerbation | 0.26 [0.22 to 0.31] | 0.38 [0.32 to 0.45] | 0.33 [0.28 to 0.39] | 0.41 [0.35 to 0.48] | 0.45 [0.39 to 0.53]
  All (mild, moderate, severe) asthma exacerbation: number analyzed (Participants) | 615 | 615 | 611 | 607 | 612
  All (mild, moderate, severe) asthma exacerbation | 0.74 [0.64 to 0.85] | 0.86 [0.75 to 0.98] | 0.93 [0.82 to 1.06] | 0.98 [0.86 to 1.11] | 1.23 [1.08 to 1.39]
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.120, Generalized linear model; Rate ratio = 0.85, 95% CI 2-sided [0.68 to 1.04]
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, Generalized linear model; Rate ratio = 0.64, 95% CI 2-sided [0.52 to 0.78]
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.170, Generalized linear modeñ; Rate ratio = 0.87, 95% CI 2-sided [0.71 to 1.06]
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.041, Generalized linear model; Rate ratio = 0.81, 95% CI 2-sided [0.66 to 0.99]
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Severe asthma exacerbation; Test type: Superiority; p = 0.050, Generalized linear model; Rate ratio = 0.78, 95% CI 2-sided [0.61 to 1.00]
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Severe asthma exacerbation; Test type: Superiority; p < 0.001, Generalized linear model; Rate ratio = 0.58, 95% CI 2-sided [0.45 to 0.73]
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Severe asthma exacerbation; Test type: Superiority; p = 0.531, Generalized linear model; Rate ratio = 0.93, 95% CI 2-sided [0.74 to 1.17]
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Severe asthma exacerbation; Test type: Superiority; p = 0.117, Linear generalized model; Rate ratio = 0.84, 95% CI 2-sided [0.67 to 1.05]
Statistical Analysis 9: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.016, Generalized linear model; Rate ratio = 0.79, 95% CI 2-sided [0.66 to 0.96]
Statistical Analysis 10: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p < 0.001, Generalized linear model; Rate ratio = 0.60, 95% CI 2-sided [0.50 to 0.72]
Statistical Analysis 11: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.161, Generalized linear model; Rate ratio = 0.87, 95% CI 2-sided [0.72 to 1.06]
Statistical Analysis 12: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p < 0.001, Generalized linear model; Rate ratio = 0.70, 95% CI 2-sided [0.58 to 0.84]

17. Secondary Outcome: Duration in Days of Asthma Exacerbations by Exacerbation Category
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS
Measure: Mean (Standard Deviation); unit: days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
days
  Moderate or severe asthma exacerbation | 4.5 (10.73) | 5.6 (12.87) | 6.7 (20.52) | 7.1 (17.17) | 8.1 (20.63)
  Severe asthma exacerbation | 2.8 (7.31) | 4.1 (11.18) | 4.9 (19.07) | 4.5 (10.54) | 5.8 (18.24)
  All (mild, moderate, severe) asthma exacerbation | 7.0 (16.02) | 8.1 (20.51) | 10.7 (28.70) | 9.6 (21.76) | 12.8 (29.21)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.183, van Elteren test
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Moderate or severe asthma exacerbation; Test type: Superiority; p < 0.001, van Elteren test
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.155, van Elteren test
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Moderate or severe asthma exacerbation; Test type: Superiority; p = 0.007, van Elteren test
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Severe asthma exacerbation; Test type: Superiority; p = 0.172, van Elteren test
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Severe asthma exacerbation; Test type: Superiority; p < 0.001, van Elteren test
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Severe asthma exacerbation; Test type: Superiority; p = 0.241, van Elteren test
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Severe asthma exacerbation; Test type: Superiority; p = 0.033, van Elteren test
Statistical Analysis 9: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.095, van Elteren test
Statistical Analysis 10: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p < 0.001, van Elteren test
Statistical Analysis 11: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p = 0.090, van Elteren test
Statistical Analysis 12: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; All (mild, moderate, severe) asthma exacerbation; Test type: Superiority; p < 0.001, van Elteren test

18. Secondary Outcome: Percentage of Participants With at Least One Asthma Exacerbation by Exacerbation Category
Description: The exacerbation categories were: All (mild, moderate and severe) and combination of moderate or severe and severe.
Time Frame: Up to Week 52
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
percentage of participants
  Moderate or severe asthma exacerbation: number analyzed (Participants) | 615 | 615 | 611 | 607 | 612
  Moderate or severe asthma exacerbation | 30.2 | 32.5 | 31.8 | 35.9 | 39.7
  Severe asthma exacerbation: number analyzed (Participants) | 615 | 615 | 611 | 607 | 612
  Severe asthma exacerbation | 21.8 | 24.6 | 23.2 | 27.3 | 29.7
  All (mild, moderate, severe) asthma exacerbation: number analyzed (Participants) | 615 | 615 | 611 | 607 | 612
  All (mild, moderate, severe) asthma exacerbation | 40.2 | 40.2 | 41.9 | 44.0 | 50.5

19. Secondary Outcome: Time in Days to Permanent Discontinuation of Study Medication Due to Asthma Exacerbation
Description: Time from start of treatment until the first event (permanent discontinuation of study medication due to asthma exacerbation) or censoring. Patients without the event were considered as censored at the date of last treatment + 1 day. For patients having the event, the date of the discontinuation of study medication was considered to calculate the time to event.
Time Frame: 52 weeks on average, up to 416 days
Population: FAS
Measure: Median (Full Range); unit: days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
days | 367.0 [11 to 416] | 367.0 [2 to 399] | 367.0 [3 to 411] | 367.0 [2 to 408] | 367.0 [2 to 416]
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p = 0.314, Regression, Cox; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.12 to 1.96]
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.055, Regression, Cox; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.08 to 1.03]
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.306, Regression, Cox; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.25 to 1.54]
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.566, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.30 to 1.94]

20. Secondary Outcome: Total Amount of Oral Corticosteroid Used (in Prednisone-equivalent mg Doses) to Treat Asthma Exacerbations
Description: The treatment of asthma exacerbations including the initiation of systemic corticosteroids were done according to investigator's or treating physician's medical judgement and in line with national and international recommendations. If systemic corticosteroids were required, a participant could return to the study after successfully completing a taper of approximately 7-10 days.
Time Frame: Up to Week 52
Population: FAS
Measure: Mean (Standard Deviation); unit: prednisone-equivalent milligram
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 615 | 616 | 611 | 607 | 612
prednisone-equivalent milligram | 53.4 (169.76) | 72.0 (211.41) | 73.2 (235.90) | 82.5 (208.36) | 86.0 (199.79)

21. Secondary Outcome: Change From Baseline in Percentage of Rescue Medication Free Days Over 26 and 52 Weeks
Description: All participants were given salbutamol/albuterol to use as rescue medication throughout the study along with e-Diary to record rescue medication use. Rescue medication free days is defined as any day where the participant did not use any puffs of rescue medication during daytime and night-time.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 590 | 577 | 578 | 580 | 579
Percentage of days
  Week 26 | 22.5 (1.32) | 19.5 (1.33) | 23.3 (1.33) | 18.2 (1.33) | 19.6 (1.33)
  Week 52: number analyzed (Participants) | 583 | 574 | 576 | 576 | 578
  Week 52 | 25.0 (1.36) | 21.9 (1.36) | 24.9 (1.36) | 20.8 (1.37) | 21.8 (1.36)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 26; Test type: Superiority; p = 0.645, LMM; LS Mean = -0.8, 95% CI 2-sided [-4.2 to 2.6], Standard Error of Mean 1.74
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.095, LMM; LS Mean = 2.9, 95% CI 2-sided [-0.5 to 6.3], Standard Error of Mean 1.73
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 26; Test type: Superiority; p = 0.460, LMM; LMM = 1.3, 95% CI 2-sided [-2.1 to 4.7], Standard Error of Mean 1.75
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 26; Test type: Superiority; p = 0.971, LMM; LS Mean = -0.1, 95% CI 2-sided [-3.5 to 3.4], Standard Error of Mean 1.75
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 52; Test type: Superiority; p = 0.963, LMM; LMM = 0.1, 95% CI 2-sided [-3.4 to 3.6], Standard Error of Mean 1.78
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.075, LMM; LS Mean = 3.2, 95% CI 2-sided [-0.3 to 6.6], Standard Error of Mean 1.77
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 52; Test type: Superiority; p = 0.517, LMM; LS Mean = 1.2, 95% CI 2-sided [-2.3 to 4.7], Standard Error of Mean 1.79
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 52; Test type: Superiority; p = 0.956, LMM; LS Mean = 0.1, 95% CI 2-sided [-3.4 to 3.6], Standard Error of Mean 1.78

22. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) at Week 52
Description: AQLQ is a 32-item disease specific questionnaire designed to measure functional impairments that are most important to patients with asthma, with a recall time of two weeks and each question to be answered on a 7-point scale (1-totally limited/problems all the time, 7-not at all limited/no problems). It consists of 4 domains:
  * Symptoms = Mean of Items 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 29, 30 (12 items)
  * Activity limitation = Mean of Items 1, 2, 3, 4, 5, 11, 19, 25, 28, 31, 32 (11 items)
  * Emotional function = Mean of Items 7, 13, 15, 21, 27 (5 items)
  * Environmental stimuli = Mean of Items 9, 17, 23, 26 (4 items)
  * Overall Score = Mean of Items 1 to 32 (32 items) The overall AQLQ score reported below is the mean of all 32 responses and ranges from 1 to 7, where higher scores indicate better quality of life.
Time Frame: 52 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 606 | 593 | 595 | 599 | 594
Score on a scale | 5.555 (0.0354) | 5.445 (0.0358) | 5.535 (0.0356) | 5.499 (0.0358) | 5.495 (0.0357)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Test type: Superiority; p = 0.690, MMRM; LS Mean = 0.020, 95% CI 2-sided [-0.078 to 0.118], Standard Error of Mean 0.0502
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.232, MMRM; LS Mean = 0.060, 95% CI 2-sided [-0.038 to 0.159], Standard Error of Mean 0.0502
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Test type: Superiority; p = 0.285, MMRM; LS Mean = -0.054, 95% CI 2-sided [-0.153 to 0.045], Standard Error of Mean 0.0506
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Test type: Superiority; p = 0.319, MMRM; LS Mean = -0.050, 95% CI 2-sided [-0.150 to 0.049], Standard Error of Mean 0.0505

23. Secondary Outcome: Pre-dose FEV1 at Weeks 4 and 12
Description: Pre-dose FEV1 is defined as average of the two FEV1 measurements taken 45 min and 15 min pre evening dose. It was assessed by performing spirometric assessment. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Time Frame: 4 weeks, 12 weeks
Population: FAS including patients with a valid measurement for the outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: litres
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 606 | 594 | 592 | 596 | 598
litres
  Week 4: number analyzed (Participants) | 598 | 573 | 573 | 579 | 577
  Week 4 | 2.032 (0.0122) | 1.983 (0.0123) | 1.963 (0.0124) | 1.950 (0.0123) | 1.887 (0.0123)
  Week 12: number analyzed (Participants) | 580 | 569 | 573 | 562 | 568
  Week 12 | 2.024 (0.0134) | 1.994 (0.0135) | 1.966 (0.0135) | 1.944 (0.0136) | 1.907 (0.0135)
Statistical Analysis 1: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.068, 95% CI 2-sided [0.036 to 0.101], Standard Error of Mean 0.0166
Statistical Analysis 2: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.145, 95% CI 2-sided [0.113 to 0.177], Standard Error of Mean 0.0165
Statistical Analysis 3: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 4; Test type: Superiority; p = 0.049, MMRM; LS Mean = 0.033, 95% CI 2-sided [0.000 to 0.066], Standard Error of Mean 0.0167
Statistical Analysis 4: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 4; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.096, 95% CI 2-sided [0.064 to 0.129], Standard Error of Mean 0.0166
Statistical Analysis 5: Comparison: QVM149 150/50/160 µg o.d. vs QMF149 150/320 µg o.d; Week 12; Test type: Superiority; p = 0.002, MMRM; LS Mean = 0.058, 95% CI 2-sided [0.022 to 0.094], Standard Error of Mean 0.0184
Statistical Analysis 6: Comparison: QVM149 150/50/160 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 12; Test type: Superiority; p < 0.001, MMRM; LS Mean = 0.117, 95% CI 2-sided [0.081 to 0.153], Standard Error of Mean 0.0183
Statistical Analysis 7: Comparison: QVM149 150/50/80 µg o.d. vs QMF149 150/160 µg o.d; Week 12; Test type: Superiority; p = 0.007, MMRM; LS Mean = 0.050, 95% CI 2-sided [0.013 to 0.086], Standard Error of Mean 0.0185
Statistical Analysis 8: Comparison: QVM149 150/50/80 µg o.d. vs Salmeterol/Fluticasone 50/500 μg b.i.d; Week 12; Test type: Superiority; p < 0.001, MMRM; MMRM = 0.087, 95% CI 2-sided [0.051 to 0.123], Standard Error of Mean 0.0184

24. Secondary Outcome: Percentage of Participants With Composite Endpoint of Serious Asthma Outcomes
Description: A composite endpoint of serious asthma outcomes is defined as asthma-related hospitalization, asthma-related intubation, or asthma-related death and was reviewed by the Adjudication Committee.
Time Frame: Up to Week 52
Population: SAF
Measure: Number; unit: Percentage of participants
Arm/Group | QVM149 150/50/160 µg o.d. | QVM149 150/50/80 µg o.d. | QMF149 150/320 µg o.d. | QMF149 150/160 µg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
Number analyzed (Participants) | 616 | 617 | 613 | 608 | 618
Percentage of participants | 1.4 | 2.5 | 1.9 | 1.6 | 1.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days (52 weeks on average, up to 416 days).
Description: Any signs or symptoms that occurs during study treatment plus the 30 days post treatment.
Groups:
- QVM149 150/50/160 μg o.d.: QVM149 150/50/160 μg (indacaterol acetate/glycopyrronium/mometasone furoate) once daily (o.d.) delivered via Concept1 device
- QVM149 150/50/80 μg o.d.: QVM149 150/50/80 μg (indacaterol acetate/glycopyrronium/mometasone furoate) once daily (o.d.) delivered via Concept1 device
- QMF149 150/320 μg o.d.: QMF149 150/320 μg (indacaterol acetate/mometasone furoate) once daily (o.d.) delivered via Concept1 device
- QMF149 150/160 μg o.d.: QMF149 150/160 μg (indacaterol acetate/mometasone furoate) once daily (o.d.) delivered via Concept1 device
Arm/Group | QVM149 150/50/160 μg o.d. | QVM149 150/50/80 μg o.d. | QMF149 150/320 μg o.d. | QMF149 150/160 μg o.d. | Salmeterol/Fluticasone 50/500 μg b.i.d.
All-Cause Mortality (participants affected / at risk) | 2/616 | 1/617 | 4/613 | 0/608 | 0/618
Serious Adverse Events (participants affected / at risk) | 46/616 | 49/617 | 52/613 | 38/608 | 39/618
Other Adverse Events (participants affected / at risk) | 367/616 | 387/617 | 377/613 | 392/608 | 419/618
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 150/50/160 μg o.d. (N=616) | QVM149 150/50/80 μg o.d. (N=617) | QMF149 150/320 μg o.d. (N=613) | QMF149 150/160 μg o.d. (N=608) | Salmeterol/Fluticasone 50/500 μg b.i.d. (N=618)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute cardiac event (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 2 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Primary biliary cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Steatohepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Bursitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Dengue fever (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
HIV infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 3 | 1 | 2
Mastoiditis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 1 | 3 | 5
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Salpingitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 2 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Alcoholic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 12 | 8 | 9
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Angiopathy (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Aortic dissection rupture (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 1 | 0
Haemorrhagic vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 2 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 150/50/160 μg o.d. (N=616) | QVM149 150/50/80 μg o.d. (N=617) | QMF149 150/320 μg o.d. (N=613) | QMF149 150/160 μg o.d. (N=608) | Salmeterol/Fluticasone 50/500 μg b.i.d. (N=618)
Pyrexia (General disorders) | 17 | 11 | 10 | 10 | 15
Bronchitis (Infections and infestations) | 49 | 48 | 46 | 44 | 55
Influenza (Infections and infestations) | 19 | 21 | 23 | 26 | 25
Lower respiratory tract infection (Infections and infestations) | 13 | 12 | 12 | 17 | 22
Nasopharyngitis (Infections and infestations) | 64 | 76 | 73 | 64 | 83
Pharyngitis (Infections and infestations) | 22 | 21 | 20 | 19 | 20
Respiratory tract infection viral (Infections and infestations) | 18 | 17 | 11 | 29 | 22
Rhinitis (Infections and infestations) | 12 | 20 | 17 | 20 | 11
Sinusitis (Infections and infestations) | 14 | 18 | 9 | 17 | 14
Upper respiratory tract infection (Infections and infestations) | 33 | 45 | 52 | 48 | 52
Upper respiratory tract infection bacterial (Infections and infestations) | 17 | 22 | 27 | 28 | 29
Urinary tract infection (Infections and infestations) | 8 | 5 | 10 | 9 | 13
Viral upper respiratory tract infection (Infections and infestations) | 21 | 31 | 38 | 26 | 47
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 14 | 5 | 12 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 18 | 18 | 16 | 14
Headache (Nervous system disorders) | 23 | 30 | 24 | 34 | 25
Asthma (Respiratory, thoracic and mediastinal disorders) | 243 | 242 | 249 | 265 | 306
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 18 | 11 | 14 | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 24 | 13 | 10 | 9 | 12
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 19 | 17 | 9 | 15 | 20
Hypertension (Vascular disorders) | 16 | 19 | 14 | 17 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT02571777/SAP_000.pdf
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT02571777/Prot_001.pdf